CLINICAL TRIAL: NCT00962221
Title: Atherogenic Lipoprotein Phenotype and LDL Size and Subclasses in Patients With Subclinical Hypothyroidism
Brief Title: Lipids Profile in Subclinical Hypothyroidism
Acronym: LPSH
Status: Terminated | Type: Observational
Why Stopped: Recruiting difficulties
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: University of Palermo (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, avraham ishay, MD, HaEmek Medical Center, Israel
Other Study IDs: 0099.09EMC
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Subclinical Hypothyroidism
Keywords: LDL lipoprotein subclasses in subclinical hypothyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- subclinical hypothyroidism: Patients with subclinical hypothyroidism
  Interventions: Procedure: laboratory analysis

INTERVENTIONS:
Procedure: laboratory analysis — laboratory analysis

SUMMARY:
Overt hypothyroidism is associated with increased risk for cardiovascular disease (CVD) as indicated by hypertension, hypercholesterolemia, and increased low-density lipoprotein cholesterol (LDL-C) levels. Mild hypothyroidism, also called subclinical hypothyroidism [SH] is highly prevalent in elderly subjects, especially in women older than 50 years of age. Whether SH is related as a risk for premature CVD is controversial. It was shown that SH is associated with elevated lipids levels, particularly LDL-cholesterol. However recent evidence suggests that the 'quality' rather than only the 'quantity' of LDL-cholesterol exerts a direct influence on the cardiovascular risk. LDL-cholesterol comprises multiple distinct subclasses that differ in their atherogenic potential. Thus, the proposed study protocol is intended to evaluate the different LDL lipoproteins subclasses in patients with subclinical hypothyroidism.

DETAILED DESCRIPTION:
Overt hypothyroidism is associated with increased risk for cardiovascular disease[CVD] as indicated by hypertension, hypercholesterolemia, and increased low-density lipoprotein cholesterol (LDL-C) levels.However, not all patients have hypertension or abnormal lipid profiles, suggesting that other factors may be involved as collagen-induced platelet aggregation or relaxation of vascular smooth muscle, elevated plasma homocysteine and C- reactive protein [CRP] levels have been reported in overt hypothyroidism and have been proposed as an independent risk factor for CVD.

Subclinical hypothyroidism [SH] is highly prevalent in elderly subjects, especially in women older than 50 years of age. Whether SH is related as a risk for premature CVD is controversial. Previously, we have demonstrated that SH in middle-aged women is associated with hypertension, hypertriglyceridemia, and elevated total cholesterol/HDL- cholesterol ratio.SH was associated with elevated plasma total cholesterol and LDL-cholesterol, decreased LDL-cholesterol/LDL-triglycerides due to decreased hepatic lipase activity. The influence of SH on lipids was directly proportional to the degree of TSH elevation.

Atherosclerosis is a diffuse disease formerly considered lipid storage disease, actually involves an ongoing inflammatory response. Elevated circulating levels of acute phase proteins, cytokines, and cell adhesion molecules indicate that inflammatory processes are occurring systematically. Metabolic syndrome is a collection of metabolic risk factors, probably of more than one cause, that appear to promote the development of atherosclerotic CVD. Hypertension, dyslipidemia and hyperglycemia are the most widely recognized characteristics of the metabolic syndrome. Individuals with metabolic syndrome manifest a prothrombotic state as well as a proinflammatory state. Insulin resistance is recognized as a chronic low-level inflammatory state. Insulin action is an important effector mechanism of the proinflammatory cytokines in CVD. Insulin resistance was proposed as the common preceding factor of hypertension, LDL and HDL-cholesterol, hypertriglyceridemia, abdominal obesity and altered glucose metabolism, linking all of these to the development of CVD. Thus, inflammation, metabolic syndrome and insulin resistance are strongly associated and play an important role in the pathogenesis of atherosclerosis. In a cross-sectional analysis, subjects with SH had a significantly higher prevalence of CVD than euthyroid subjects. There were more cardiovascular deaths in subjects with SH than in the euthyroid population. These data suggest that SH may be an independent risk factor for CVD. It is not clear yet whether patients with SH have cardiovascular risk, as do patients with overt hypothyroidism, and whether metabolic syndrome and insulin resistance already exist in untreated patients with SH.

This question was recently studied by our group. We evaluated untreated patients with SH. the percentage of MS in patients (41.5%) was significantly higher than in controls (12.2%; p=0.003]. SH had significantly higher likelihood of cardiovascular risks [odds ratio 6.26, 95% confidence interval (CI) 1.6 - 4.49, p= 0.008 for MS].

We conclude that SH is associated with greater probability of MS. Recent evidence suggests that the 'quality' rather than only the 'quantity' of LDL exerts a direct influence on the cardiovascular risk. LDL comprises multiple distinct subclasses that differ in size, density, physicochemical composition, metabolic behaviour and atherogenicity. There are at least four major subspecies of LDL (e.g. large LDL-I, medium LDL-II, small LDL-III, very small LDL-IV) and the predominance of small dense LDL has been accepted as an emerging cardiovascular risk factor.

Thus, the proposed study protocol is intended to evaluate lipoprotein phenotype and LDL size and subclasses in patients with subclinical Hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with subclinical hypothyroidism

Exclusion Criteria:

* Patients taking L-thyroxin therapy
* Patients with known cardiovascular, cerebral or peripheral atherosclerotic disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at the Endocrine Institute, Haemek Medical Center, Afula, Israel
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of atherogenic lipoproteins | enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Luboshitzky, MD, Study Director — Endocrine Institute, Haemek Medical Center, Afula, Israel; Manfredi Rizzo, MD, Study Chair — University of Palermo; Giatgen Spinas, MD, Study Chair — University of Zurich; Kaspar Berneis, MD, Study Chair — University of Zurich
Locations (1):
- Endocrine Institute, Haemek Medical Center, Afula, Israel